CLINICAL TRIAL: NCT05383937
Title: Comparative Impact of Protocolized Management, Intensive Rehabilitation Versus Long-term Classic Rehabilitation of Dyslexic Children.
Acronym: INTENS-DYS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitement diffculties
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/692
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dyslexia; Speech Therapy; Children, Only
Keywords: Dyslexia; Speech Therapy; Children; Intensive rehabilitation
MeSH Terms: conditions — Dyslexia; Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive arm (Experimental): The children included in this arm will receive two weeks of daily care during which two daily speech therapy sessions of one hour each will be performed. This will be done between M2 and M4 of inclusion in order to avoid potential measurement bias. These sessions will be carried out by a state-qualified speech therapist employed at the CRRF of Bregille. They will guide the intensive rehabilitation of dyslexic children by focusing the exercises on their main difficulties.
  Interventions: Other: Speech Therapy INTENS-DYS
- classic arm or gold standard (Active Comparator): The speech therapy session will be provided only by private practitioners, with a weekly consultation of 30 minutes. The private speech therapist who initially referred the patient for inclusion in the research protocol will be responsible for his or her "classic" rehabilitation. The therapy will continue during the 6 months of research.
  Interventions: Other: Speech Therapy INTENS-DYS

INTERVENTIONS:
Other: Speech Therapy INTENS-DYS — During the six research month, children included in the intensive arm will benefit of two daily hours speech therapy during two weeks. Those one will be carried out between the second and the fourth month.

SUMMARY:
Dyslexia is characterized by difficulties with accurate and/or fluent word recognition and by poor spelling and decoding abilities. In France, dyslexia is a public health disorder. Dyslexia is a real public health problem in France, affecting 6% of the general population. However, no clinical trial of a standardized rehabilitation has shown an impact on reading fluency. In the era of intensive rehabilitation, a new protocol based on the current data from the medical literature has been designed.

ELIGIBILITY:
Inclusion Criteria:

* Children from 8 to 12 years old,
* Living in and around 50 kilometers from Besançon.
* Diagnosis of dyslexia according to the DSM-V or CIM-10 requirements.
* Consent form signed by the parental authority and the child,
* Affiliation to a social security system.

Exclusion Criteria:

* Mother's medical history of pregnancy or delivery complications,
* Patients's medical history of neurological infectious, vascular or tumoral events,
* Patient's medical history of intellectual deficiency,
* Patients's medical history of visual or hearing disorders,
* Patient's medical history of psychiatric disorders (especially diagnosis of Attention Deficit / Hyperactivity Disorders (AD/HD)),
* legal incapacity,
* limited cooperation suspected by the investigator.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Reading fluency to the Alouette test. | Six month.
  Difference in the number of words read correctly in three minutes in the intensive and the conventional arm.

SECONDARY OUTCOMES:
Phonological processing tests. | Six month.
  Difference in the number of errors in logatom repetition, which means phonological rules of a language corresponding of meaningless words, in the intensive and the conventional arm.
Visual pattern. | Six month.
  Difference in the number of errors to five visual pattern from the BALE and the EVALEO, in the intensive and the conventional arm.
Life Quality. | 6 month.
  Difference on the AUQUEI self questionnary, in the intensive and the conventional arm.
Rehabilitation adhesion. | 6 month
  Number of speech therapy session performed by patient in each arms.
Speech langage rehabilitation cost. | 6 month.
  Differential cost/progress relation of intensive and classical rehabilitation.
Family and school evaluation. | 6 month.
  Difference to Visual Analog Scale (VAS) regarding the benefit of speech therapy rehabilitation, assessed by the family and the school teachers, in each arms.

CONTACTS AND LOCATIONS:
Overall Officials: Julien BEVALOT, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No